CLINICAL TRIAL: NCT06804603
Title: A Proof of Concept, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of Tradipitant on Nausea and Vomiting After GLP-1R Agonist Administration in Healthy Overweight Class I or Class II Obese Volunteers
Brief Title: A Study to Measure the Effects of Using Tradipitant on Nausea and Vomiting After GLP-1R Agonist Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VLY-686-2601
Record Dates: First submitted 2025-01-09; First posted 2025-02-03 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: GLP-1R agonist; semaglutide; obesity; nausea; vomiting
MeSH Terms: conditions — Obesity; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Treatment with placebo BID for approximately 2 weeks
  Interventions: Drug: Placebo
- Tradipitant Group (Experimental): Treatment with tradipitant BID for approximately 2 weeks
  Interventions: Drug: Tradipitant

INTERVENTIONS:
Drug: Tradipitant — Oral capsule
  Arms: Tradipitant Group
Drug: Placebo — Oral capsule
  Arms: Placebo Group

SUMMARY:
The goal of this study is to measure the effects of using Tradipitant after GLP-1R agonist use on nausea and vomiting in healthy overweight, class I, or class II obese volunteers. The study is placebo-controlled with two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index 25-40 kg/m^2 inclusive
* No serious medical problems or chronic diseases, specifically no type I or type II diabetes

Exclusion Criteria:

* Another disorder that contributes to gastrointestinal symptoms
* History of intolerance and/or hypersensitivity to NK-1 receptor antagonists
* History of intolerance and/or hypersensitivity to GLP-1 receptor agonists
* Exposure to any investigational medication within the past 60 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with at least 1 vomiting episode per week in the tradipitant group compared to the placebo group as measured by a daily symptom diary. | 1 week
  A daily diary called the Nausea Vomiting Daily Diary (NV-DD) will be used. The NV-DD asks participants to rate their nausea symptoms on a Likert scale from 0-5 (0=none, 5= very severe), as well as record the duration of nausea and vomiting frequency.

SECONDARY OUTCOMES:
Individual gastrointestinal symptoms | 1 week
  Nausea and vomiting symptoms will be assessed using the NV-DD. The NV-DD asks participants to rate their nausea symptoms on a Likert scale from 0-5 (0=none, 5= very severe), as well as record the duration of nausea and vomiting frequency.
Safety and tolerability of tradipitant after administration of semaglutide as measured by spontaneous reporting of adverse events (AEs) | 2 weeks
  Safety will be monitored using vital signs, blood chemistry, hematology, urology, and ECGs (QT, PR, QTcF, QTcB, QRS intervals and heart rate).

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (3):
- United States (3):
  - Vanda Investigational Site, Los Angeles, California
  - Vanda Investigational Site, Rochester, Minnesota
  - Vanda Investigational Site, New York, New York

IPD SHARING:
Plan to Share IPD: No